CLINICAL TRIAL: NCT02201979
Title: Laser Fluorescent Imaging of Nipple and Areola During Breast Lift in Combination With Breast Implants
Brief Title: Laser Fluorescent Imaging of Nipple and Areola During Breast Lift
Status: Completed | Type: Observational
Sponsor: Swanson Center (Other)
Responsible Party: Principal Investigator, Eric Swanson, M.D., Principal Investigator, Swanson Center
Other Study IDs: Swanson 004
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Breast Sagging; Ptosis; Loss of Breast Volume
Keywords: breast; ptosis; sagging; implant; lift
MeSH Terms: conditions — Blepharoptosis | interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast lift in combination with implants.: Patients undergoing breast lifts in combination with implants are studied using laser fluorescent imaging to evaluate blood supply.
  Interventions: Procedure: Vertical breast lift with implants

INTERVENTIONS:
Procedure: Vertical breast lift with implants

SUMMARY:
Breast lift surgery performed in combination with breast implants is a common cosmetic operation. However, there have been concerns regarding the safety of this treatment combination. Some investigators are concerned that an implant may increase the risk of complications, including loss of circulation to the nipple and areola. This study was undertaken to evaluate the blood supply of the breast using intraoperative laser fluorescent imaging and to determine whether a breast implant compromises blood supply to the nipple and areola.

DETAILED DESCRIPTION:
Protocol

Laser Fluorescent Imaging of Breasts During Vertical Breast Lifts and Reductions Performed in Combination with Breast Implants.

Background/Purpose

Today, breast lifts are a common operation. Implants may be recommended to provide greater fullness of the upper poles of the breasts. One of the risks of surgery is compromised circulation to the nipples and areolae. Some investigators believe that the simultaneous insertion of breast implants adds to the risk by causing pressure on the overlying breast tissue and skin.1 Staging the procedure (first the breast lift and then implants or vice versa) has been recommended, but staging is inconvenient and costly for patients, necessitating two operations. Clinical experience with the newer vertical breast lift technique, as opposed to the traditional inferior pedicle technique, has been favorable, with few reported complications.2 The vertical technique uses a shorter, more superficial pedicle than the traditional inferior pedicle, with a more reliable blood supply.2 A breast lift and reduction are essentially the same operation; more breast tissue is removed during a reduction but the dissection is the same.

This study was undertaken to investigate the blood supply to the nipples and areolae during the combined breast lift/reduction and implants procedure. Laser fluorescent imaging represents an objective measurement technique that has been used for several years to monitor the vascularity of flaps used in breast reconstruction.

Subjects

Fifteen consecutive consenting adult women undergoing outpatient elective breast lifts or reductions in combination with breast implants will be investigated. By testing the blood supply at two time points, the patient serves as her own control.

Imaging

The SPY Elite Intraoperative Perfusion Assessment System (Lifecell Corp., Branchburg, NJ) consists of a near-infrared laser that detects fluorescence. The imaging agent, indocyanine green, is absorbed at 800-810 nm. The imaging agent is injected intravenously. Starting within 5-10 seconds of injection, the system records images of the breasts, showing the fluorescence, which indicates blood supply. The half-life of the imaging agent is 2.5-3 minutes.

Surgery

The implants are inserted and the breast lift/reduction procedure is performed on both sides using the vertical technique.2 The implants are not inflated. The filling tubes are left in place. At this point, 3 mL (7.5 mg) of indocyanine green is injected and the image is recorded, documenting blood supply to both breasts. Next, the implants are inflated using the filling tubes. After inflation of the implants, the breasts are reimaged, with the filling tubes still in place. Once adequate circulation is demonstrated, the filling tubes are removed. In the unlikely event that inadequate circulation is found during imaging, the implant volume may be reduced accordingly, and a third image taken to confirm adequate circulation to the nipples.

Null Hypothesis

A breast lift or reduction performed using the vertical technique in combination with insertion of breast implants does not compromise circulation to the nipples and areolae and may be safely performed simultaneously, avoiding a need for staged surgery.

Informed Consent

Patients are informed as to the nature of the study and are told that their participation is entirely voluntary and they are free to decline, and that doing so does not in any way prejudice their treatment. Patients are informed of the small risk of an allergic reaction that will be treated if it occurs.

Patient Risk

There is no patient risk apart from a very small risk of allergic reaction, which is further reduced by excluding any patient with a known allergy to iodinated contrast dye. The study does not affect patient treatment. It offers the possibility of detection of reduced skin circulation, information that can be used by the surgeon to limit implant volume, or forego their simultaneous insertion if necessary and reduce the risk of tissue loss and delayed wound healing, known complications of breast lifts and reductions.

Sample Size

A sample of 15 patients is anticipated, treated over a period of approximately 5 months.

Disclosure

The author has no financial interest in any of the products, devices, or drugs mentioned in this article. The author has no conflicts of interest to disclose. There was no outside funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 80
* Consent for participation

Exclusion Criteria:

* history of allergy to iodinated contrast dye -

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women undergoing cosmetic breast lifts in combination with implants.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Blood supply to breast as evaluated by laser fluorescent imaging | 5 months
  Laser fluorescent imaging is used to evaluate breast blood supply.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swanson, M.D., Principal Investigator — Swanson Center
Locations (1):
- Swanson Center, Leawood, Kansas, United States

REFERENCES:
- [Background] Swanson E. Prospective comparative clinical evaluation of 784 consecutive cases of breast augmentation and vertical mammaplasty, performed individually and in combination. Plast Reconstr Surg. 2013 Jul;132(1):30e-45e. doi: 10.1097/PRS.0b013e3182910b2e. PMID 23806952